CLINICAL TRIAL: NCT00681434
Title: Bilateral Training for Upper Extremity Hemiparesis in Stroke
Brief Title: Bilateral Training Versus Unilateral Training in Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Shirley Ryan AbilityLab (Other)
Responsible Party: Daniel M. Corcos, PhD, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006-0234
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Stroke; Hemiparesis
Keywords: stroke; upper extremity; hemiparesis
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): bilateral training
  Interventions: Behavioral: bilateral upper extremity training
- 2 (Active Comparator): Unilateral training
  Interventions: Behavioral: Unilateral upper extremity training

INTERVENTIONS:
Behavioral: bilateral upper extremity training — Bilateral symmetrical upper extremity training for proximal control for three hours per week for eight weeks.
  Arms: 1
Behavioral: Unilateral upper extremity training — Unilateral upper extremity training for proximal extremity for three hours a week for eight weeks.
  Arms: 2

SUMMARY:
This randomized, single-blind study compares the effectiveness of bilateral training to unilateral training for individuals with moderate hemiparesis. We hypothesize that bilateral training will be superior to unilateral in the proximal extremity but not the distal one.

DETAILED DESCRIPTION:
Upper extremity hemiparesis is the most common post-stroke disability. Longitudinal studies have indicated that 30 to 66 percent of stroke survivors do not have full arm function six months post-stroke. Bilateral arm training has been investigated as a potential rehabilitation intervention for individuals not eligible for constraint induced movement therapy.

This training study included 24 hours of treatment over eight weeks. The protocol consisted of reaching activities with rhythmic auditory cueing emphasizing the proximal arm. Subjects assigned to the bilateral group performed bilateral symmetrical activities while subjects in the unilateral group performed the same activity with the affected arm only. The Motor Assessment Scale-Upper Limb Item and the Motor Status Scale are used as primary outcome measures. The Reaching Performance Scale and strength measures are secondary outcome measures. Assessments are administered pre-/ and post-training by a blind rater.

ELIGIBILITY:
Inclusion Criteria:

* cortical or subcortical stroke
* chronic condition (at least six months prior)
* ability to follow 2-step commands
* ability to give consent

Exclusion Criteria:

* lesion in brain stem or cerebellum
* visual field cut
* neglect
* uncontrolled hypertension
* angina
* COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-05; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Motor Assessment Scale | pre and post (week one and week 8)
Motor Status Scale | pre and post, Week 0 and Week eight

SECONDARY OUTCOMES:
Reaching Performance Scale | pre and post training (Week 0 and week 8)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Stoykov, PhD, Principal Investigator — University of Illinois at Chicago Department of Kinesiology and Nutrition; Daniel M Corcos, PhD, Study Chair — University of Illinois at Chicago Department of Kinesiology and Nutrition

REFERENCES:
- [Result] Stoykov ME, Lewis GN, Corcos DM. Comparison of bilateral and unilateral training for upper extremity hemiparesis in stroke. Neurorehabil Neural Repair. 2009 Nov;23(9):945-53. doi: 10.1177/1545968309338190. Epub 2009 Jun 16. PMID 19531608